CLINICAL TRIAL: NCT05381948
Title: A Phase 2, Multicenter, Prospective, Randomized, Double-Masked, Parallel Study of EYP-1901, a Tyrosine Kinase Inhibitor (TKI), Compared to Aflibercept in Subjects With Wet AMD
Brief Title: Study of EYP-1901 in Subjects With Wet Age Related Macular Degeneration (wAMD)
Acronym: DAVIO2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EYP-1901-201
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: wAMD; EYP-1901; EyePoint
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EYP-1901 2060 mcg (Experimental): EYP-1901 2060 mcg, single dose
  Interventions: Drug: EYP-1901
- EYP-1901 3090 mcg (Experimental): EYP-1901 3090 mcg, single dose
  Interventions: Drug: EYP-1901
- Aflibercept (Active Comparator): Aflibercept 2 milligram (mg) [0.05 milliliter (mL)] every 8 weeks
  Interventions: Drug: Aflibercept 2mg/0.05mL Inj,Oph

INTERVENTIONS:
Drug: EYP-1901 — Intravitreal Injection
  Arms: EYP-1901 2060 mcg; EYP-1901 3090 mcg
Drug: Aflibercept 2mg/0.05mL Inj,Oph — Intravitreal Injection
  Other Names: Eylea
  Arms: Aflibercept

SUMMARY:
This is a phase 2 randomized, double -masked study comparing the efficacy of EYP-1901 at 2 dose levels: 2060 microgram (mcg) and 3090 mcg against aflibercept.

DETAILED DESCRIPTION:
This study is evaluating the 2 doses of EYP-1901 against aflibercept in a randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of wAMD in the study eye, with disease onset any time prior to the Screening Visit.
* Documented anatomical response (that is, reduction in fluid on [spectral-domain - optical coherence tomography (SD-OCT)] to previous intravitreal anti-vascular endothelial growth factor (anti-VEGF) injections in the study eye prior to the Screening Visit.
* Previously treated with at least 2 anti-VEGF intravitreal injections (that is, bevacizumab, ranibizumab, aflibercept or faricimab) for wAMD per standard of care in the study eye within 6 months prior to the Screening Visit.
* Received previous anti-VEGF therapy 2 to 5 weeks (14 to 35 days) in the study eye prior to Screening Visit, but no more than 42 days prior to randomization to study treatment on Day 1.
* Best corrected visual acuity (BCVA) early Treatment Diabetic Retinopathy Study (ETDRS) letter score of 35 letters (20/200 Snellen equivalent) to 85 letters (20/20 Snellen equivalent) in the study eye at the Screening Visit and on Day 1.
* Able to understand, and willingness to sign, the informed consent and to provide access to personal health information via Health Insurance Portability and Accountability Act (HIPAA) authorization.
* Willingness and ability to comply with all scheduled visits, restrictions, and assessments.
* For women of childbearing potential, or men with female partners of childbearing potential, agreement to the use of an appropriate form of contraception at the Screening Visit and for the duration of the study.

Exclusion Criteria:

* History of pars plana vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in the study eye.
* Prior treatment with Visudyne® (verteporfin), external beam radiation therapy, or transpupillary thermotherapy in the study eye.
* Previous treatment with intravitreal corticosteroid injection or device implantation in the study eye.
* Previous focal laser photocoagulation used for AMD treatment in the study eye.
* Total choroidal neovascularization (CNV) lesion size >12 disc areas [30.5 millimeter square (mm^2)] as assessed by fluorescein angiography (FA) in the study eye at the Screening Visit.
* Central subfield thickness (CST) >350 micrometer (mcm) in the study eye at the Screening Visit or Day 1.
* Intraretinal cystic fluid >25 mcm in diameter involving the central subfield and/or disruption of normal morphology (loss of foveal depression, disruption of external limiting membrane) secondary to cystic intraretinal fluid within the central subfield, in the study eye at the Screening Visit. Diffuse (non-cystic) intraretinal fluid would not be excluded.
* Subretinal hemorrhage in the subfoveal/juxtafoveal location and hemorrhage greater than 1 disc are (1.8 mm^2) if located less than 200 mcm from the foveal center in the study eye at either the Screening Visit or Day 1.
* Subfoveal fibrosis, atrophy, or scarring in the center subfield in the study eye at the Screening Visit.
* Fibrosis >50% of the total lesion, in the study eye at the Screening Visit.
* Retinal pigment epithelium detachment (RPED) thickness >400 mcm at any point within 3 mm of the foveal center in the study eye at either the Screening Visit or Day 1.
* Retinal pigment epithelial tear in the study eye at the Screening Visit or Day 1.
* Any concurrent intraocular condition in the study eye (e.g., cataract or glaucoma) that, in the opinion of the investigator, would have either required surgical intervention during the study to prevent or treat visual loss that might result from that condition or affected interpretation of the study results.
* Historical or active intraocular inflammation (grade trace or above) in the study eye, other than expected findings from routine cataract surgery.
* History of vitreous hemorrhage in the study eye within 12 weeks prior to the Screening Visit.
* History of rhegmatogenous retinal detachment or treatment for retinal detachment or macular hole (stage 3 or 4) in the study eye.
* Aphakia or pseudophakia with the absence of the posterior capsule in the study eye (YAG capsulotomy is permitted).
* Spherical equivalent of the refractive error in the study eye demonstrating >8 diopters of myopia.
* For subjects who have undergone prior refractive or cataract surgery in the study eye, preoperative refractive error in the study eye exceeding 8 diopters of myopia.
* Intraocular surgery (including cataract surgery) in the study eye within 12 weeks prior to the Screening Visit.
* Uncontrolled ocular hypertension or glaucoma in the study eye (defined as intraocular pressure (IOP) >25 mm of mercury (mmHg) or a cup to disc ratio >=0.8, despite treatment with 2 or more classes of antiglaucoma medication) and any such condition which the Investigator feels may require a glaucoma-filtering surgery while in the study.
* History of glaucoma-filtering surgery, tube shunts, or microinvasive glaucoma surgery in the study eye.
* History of corneal transplant in the study eye.
* BCVA using ETDRS charts <30 letters (20/250 Snellen equivalent) in the fellow eye.
* Worsening of BCVA ≥10 ETDRS letters in the study eye from the Screening Visit to Day 1.
* Presence of CNV in either eye due to other causes aside from wAMD at the Screening Visit.
* Treatment with Visudyne® in the fellow eye <7 days prior to the Screening Visit.
* Prior participation in a clinical trial involving investigational anti-angiogenic drugs administered in either eye or systemically within 8 weeks prior to the Screening Visit.
* Prior participation in a clinical trial involving investigational ocular gene therapy trial for either eye.
* History of idiopathic or autoimmune-associated uveitis in either eye.
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye.
* Presence of any other systemic or ocular condition which, in the judgment of the investigator, could make the subject inappropriate for entry into this study.
* Uncontrolled blood pressure (defined as systolic >180 mmHg and/or diastolic >100 mmHg), based on the average of three readings taken with the subject in a resting state.
* Myocardial infarction within 6 months prior to screening or New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled atrial fibrillation, uncontrolled angina, cardiomyopathy, ventricular arrhythmias or other cardiac conditions which, in the judgment of the investigator, could make the subject inappropriate for entry into this study.
* Serious non-healing wound, ulcer, or bone fracture.
* Glycated hemoglobin (HbA1c) greater than 7% at the Screening Visit.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of EYP-1901.
* Current treatment for any active systemic infection.
* Previous use of any systemic anti-VEGF agents or intraocular brolucizumab in the study eye.
* Use of oral corticosteroids (prednisone >10 mg/day or equivalent) within 30 days prior to the Screening Visit.
* History or presence of bleeding disorders, including platelet disorders, hemorrhage, acquired or hereditary coagulation disorders (including deep vein thrombosis and pulmonary embolisms), acquired or hereditary vascular disorders, stroke, or transient ischemic attack.
* Excluding certain skin cancers (specifically, basal cell carcinoma and squamous cell carcinoma), any malignancy receiving treatment, or in remission less than 5 years prior to study entry.
* History of allergy to fluorescein, not amenable to treatment.
* Inability to obtain fundus photographs, FA, fundus autofluorescence, or SD-OCT images of sufficient quality to be analyzed and graded by the Central Reading Center.
* Historical or active diagnosis of any medical or psychological condition that could interfere with the ability of the subject to give informed consent, or to comply with study or follow-up procedures.
* Previous participation in any ocular or non-ocular (systemic) disease studies of investigational drugs within 30 days prior to the Screening Visit (excluding vitamins and minerals).
* Use of anti-mitotic or anti-metabolite therapy within 30 days or 5 elimination half-lives of the Screening Visit, whichever is longer.
* Intolerance, contraindication, or hypersensitivity to topical anesthetics, dyes, povidone iodine, mydriatic medications, or any of the ingredients of the EYP-1901 insert.
* Requirement for continuous use of any protocol-prohibited medications or treatments.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception during the study as outlined in this protocol.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-04-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (67):
- United States (67):
  - EyePoint Investigative Site, Phoenix, Arizona
  - EyePoint Investigative Site, Springdale, Arkansas
  - EyePoint Investigative Site, Beverly Hills, California
  - EyePoint Investigative Site, Campbell, California
  - EyePoint Investigative Site, Encino, California
  - EyePoint Investigative Site, Fullerton, California
  - EyePoint Investigative Site, Glendale, California
  - EyePoint Investigative Site, Huntington Beach, California
  - EyePoint Investigative Site, Irvine, California
  - EyePoint Investigative Site, Pasadena, California
  - EyePoint Investigative Site, Poway, California
  - EyePoint Investigative Site, Redlands, California
  - EyePoint Investigative Site, Sacramento, California
  - EyePoint Investigative Site, Walnut Creek, California
  - EyePoint Investigative Site, Lakewood, Colorado
  - EyePoint Investigative Site, Clearwater, Florida
  - EyePoint Investigative Site, Coral Springs, Florida
  - EyePoint Investigative Site, Lakeland, Florida
  - EyePoint Investigative Site, Melbourne, Florida
  - EyePoint Investigative Site, Miami, Florida
  - EyePoint Investigative Site, Pensacola, Florida
  - EyePoint Investigative Site, Sarasota, Florida
  - EyePoint Investigative Site, St. Petersburg, Florida
  - EyePoint Investigative Site, Tampa, Florida
  - EyePoint Investigative Site, Winter Haven, Florida
  - EyePoint Investigative Site, Marietta, Georgia
  - EyePoint Investigative Site, ‘Aiea, Hawaii
  - EyePoint Investigative Site, Chicago, Illinois
  - EyePoint Investigative Site, Lemont, Illinois
  - EyePoint Investigative Site, Carmel, Indiana
  - EyePoint Investigative Site, West Des Moines, Iowa
  - EyePoint Investigative Site, Baltimore, Maryland
  - EyePoint Investigative Site, Hagerstown, Maryland
  - EyePoint Investigative Site, Owings Mills, Maryland
  - EyePoint Investigative Site, Boston, Massachusetts
  - EyePoint Investigative Site, Springfield, Massachusetts
  - EyePoint Investigative Site, Grand Rapids, Michigan
  - EyePoint Investigative Site, Saint Louis, Michigan
  - EyePoint Investigative Site, St Louis, Missouri
  - EyePoint Investigative Site, Reno, Nevada
  - EyePoint Investigative Site, Teaneck, New Jersey
  - EyePoint Investigative Site, Great Neck, New York
  - EyePoint Investigative Site, Hauppauge, New York
  - EyePoint Investigative Site, Liverpool, New York
  - EyePoint Investigative Site, Shirley, New York
  - EyePoint Investigative Site, Asheville, North Carolina
  - EyePoint Investigative Site, Wake Forest, North Carolina
  - EyePoint Investigative Site, Eugene, Oregon
  - EyePoint Investigative Site, Portland, Oregon
  - EyePoint Investigative Site, Springfield, Oregon
  - EyePoint Investigative Site, Charleston, South Carolina
  - EyePoint Investigative Site, West Columbia, South Carolina
  - EyePoint Investigative Site, Germantown, Tennessee
  - EyePoint Investigative Site, Nashville, Tennessee
  - EyePoint Investigative Site, Abilene, Texas
  - EyePoint Investigative Sites, Austin, Texas
  - EyePoint Investigative Site, Dallas, Texas
  - EyePoint Investigative Sites, Houston, Texas
  - EyePoint Investigative Site, McAllen, Texas
  - EyePoint Investigative Site, Plano, Texas
  - EyePoint Investigative Site, San Antonio, Texas
  - EyePoint Investigative Site, The Woodlands, Texas
  - EyePoint Investigative Site, Salt Lake City, Utah
  - EyePoint Investigative Site, Fairfax, Virginia
  - EyePoint Investigative Site, Lynchburg, Virginia
  - EyePoint Investigative Site, Warrenton, Virginia
  - EyePoint Investigative Site, Silverdale, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2 prospective, randomized, double-masked study was conducted in previously treated subjects with wet age-related macular degeneration (wAMD) at 39 sites in the United States between 30 June 2022 and 24 April 2024.
Pre-assignment Details: This study consists of a screening period (up to 14 days) and treatment period (56 weeks). A total of 161 subjects were randomized in the study.
Groups:
- Aflibercept 2 mg: Subjects received aflibercept 2 mg intravitreal injection on Day 1 and at Week 4 followed by intravitreal injection of aflibercept 2 mg and sham injection at Week 8 and then aflibercept 2 mg intravitreal injection once every 8 weeks up to Week 56.
- EYP-1901 2060 mcg: Subjects received aflibercept 2 mg intravitreal injection on Day 1 and at Week 4 followed by intravitreal injection of aflibercept 2 mg and EYP-1901 2060 mcg injection at Week 8 and then intravitreal sham injection once every 8 weeks up to Week 56.
- EYP-1901 3090 mcg: Subjects received aflibercept 2 mg intravitreal injection on Day 1 and at Week 4 followed by intravitreal injection of aflibercept 2 mg and EYP-1901 3090 mcg injection at Week 8 and then intravitreal sham injection once every 8 weeks up to Week 56.
Period: Overall Study
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Started | 54 | 53 | 54
Completed | 52 | 47 | 52
Not Completed | 2 | 6 | 2
Not completed — Adverse Event: Ocular - Study Eye | 0 | 1 | 0
Not completed — Adverse Event: Non-ocular | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Deviation | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Death | 0 | 2 | 0
Not completed — Discontinued study without receiving study drug | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized subjects who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg | Total
Number analyzed (Participants) | 54 | 50 | 52 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.9 (7.59) | 76.4 (6.66) | 75.4 (7.19) | 75.9 (7.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 35 | 96
  Male | 25 | 18 | 17 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 3 | 4
  Not Hispanic or Latino | 53 | 48 | 49 | 150
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 1
  Black | 0 | 0 | 0 | 0
  White | 53 | 50 | 51 | 154
  Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Average Change in Best Corrected Visual Acuity (BCVA) From Baseline Averaged Over Weeks 28 and 32
Description: The BCVA was measured according to the standard procedure originally developed for Early Treatment Diabetic Retinopathy Study (ETDRS). The ETDRS letter score calculated when 20 or more letters were read correctly at 4.0 meters; the visual acuity letter score was equal to the total number of letters read correctly at 4.0 meters plus 30. The score ranges from 0 (worse) to 100 (best). Higher scores indicate positive outcome measure. Baseline was defined as the last non-missing measurement before the initiation of study treatment.
Time Frame: Baseline (Day 1) and Weeks 28 and 32
Population: The Full Analysis Set (FAS) included all randomized subjects who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 54 | 50 | 52
score on a scale | 1.17 (0.830) | 1.05 (0.866) | 0.87 (0.841)
Statistical Analysis 1: Comparison: Aflibercept 2 mg vs EYP-1901 2060 mcg; Test type: Other; p = 0.919, Mixed Model for Repeated Measures (MMRM); Least Square (LS) Mean = -0.12, 95% CI 2-sided [-2.48 to 2.24], Standard Error of Mean 1.199
Statistical Analysis 2: Comparison: Aflibercept 2 mg vs EYP-1901 3090 mcg; Test type: Other; p = 0.795, MMRM; LS Mean = -0.31, 95% CI 2-sided [-2.63 to 2.02], Standard Error of Mean 1.187

2. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity up to Week 56
Description: The BCVA was measured according to the standard procedure originally developed for ETDRS. The ETDRS letter score calculated when 20 or more letters were read correctly at 4.0 meters; the visual acuity letter score was equal to the total number of letters read correctly at 4.0 meters plus 30. The score ranges from 0 (worse) to 100 (best). Higher scores indicate positive outcome measure. Baseline was defined as the last non-missing measurement before the initiation of study treatment.
Time Frame: Baseline (Day 1) and Weeks 32 and 56
Population: The FAS included all randomized subjects who received at least 1 dose of study treatment. Only subjects analyzed at baseline and specific timepoints are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 54 | 50 | 52
score on a scale
  Baseline (Day 1) | 73.4 (9.48) | 73.9 (7.90) | 74.9 (7.68)
  Week 32: number analyzed (Participants) | 53 | 48 | 52
  Week 32 | 1.6 (6.81) | 1.0 (6.45) | 0.8 (5.22)
  Week 56: number analyzed (Participants) | 52 | 47 | 52
  Week 56 | 1.1 (8.55) | 0.3 (8.10) | -1.9 (7.83)

3. Secondary Outcome: Percentage of Subjects With >=5, >=10, and >=15 BCVA Letter Change From Baseline up to Week 56
Description: as for outcome 2
Time Frame: Baseline (Day 1) and Weeks 32 and 56
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 53 | 48 | 52
percentage of subjects
  Week 32: >=5 BCVA Letter Gain | 34.0 | 25.0 | 21.2
  Week 32: >=5 BCVA Letter Loss | 13.2 | 20.8 | 11.5
  Week 32: >=10 BCVA Letter Gain | 5.7 | 10.4 | 5.8
  Week 32: >=10 BCVA Letter Loss | 5.7 | 6.3 | 3.8
  Week 32: >=15 BCVA Letter Gain | 1.9 | 2.1 | 0
  Week 32: >=15 BCVA Letter Loss | 1.9 | 0 | 1.9
  Week 56: >=5 BCVA Letter Gain: number analyzed (Participants) | 52 | 47 | 52
  Week 56: >=5 BCVA Letter Gain | 32.7 | 23.4 | 15.4
  Week 56: >=5 BCVA Letter Loss: number analyzed (Participants) | 52 | 47 | 52
  Week 56: >=5 BCVA Letter Loss | 23.1 | 23.4 | 32.7
  Week 56: >=10 BCVA Letter Gain: number analyzed (Participants) | 52 | 47 | 52
  Week 56: >=10 BCVA Letter Gain | 17.3 | 12.8 | 3.8
  Week 56: >=10 BCVA Letter Loss: number analyzed (Participants) | 52 | 47 | 52
  Week 56: >=10 BCVA Letter Loss | 11.5 | 10.6 | 13.5
  Week 56: >=15 BCVA Letter Gain: number analyzed (Participants) | 52 | 47 | 52
  Week 56: >=15 BCVA Letter Gain | 1.9 | 4.3 | 0
  Week 56: >=15 BCVA Letter Loss: number analyzed (Participants) | 52 | 47 | 52
  Week 56: >=15 BCVA Letter Loss | 7.7 | 4.3 | 3.8

4. Secondary Outcome: Percentage of Subjects Not Receiving Supplemental Injection of Aflibercept up to Week 56
Description: Supplemental therapy was any unscheduled injection of aflibercept, whether or not a subject had met rescue criteria. For the aflibercept arm, any aflibercept injection following Week 8 which did not occur at Weeks 16, 24, 32, 40, 48, or 56, was supplemental therapy. For either of the EYP-1901 arms, any aflibercept injection following the Week 8 visit was supplemental therapy.
Time Frame: Weeks 32 and 56
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 53 | 48 | 52
percentage of subjects
  Week 32 | 94.3 | 62.5 | 63.5
  Week 56: number analyzed (Participants) | 52 | 47 | 52
  Week 56 | 82.7 | 42.6 | 46.2

5. Secondary Outcome: Median Time to First Supplemental Aflibercept Injection in the Study Eye Following the EYP-1901 Dose at Week 8
Description: Time to first supplemental aflibercept injection following Week 8 study treatment was defined as the date of the first supplemental aflibercept injection minus the date of the Week 8 study treatment administration, divided by 7 days per week. Subjects who did not receive any supplemental aflibercept injection following study treatment administration at Week 8 were censored at their date of last visit (those who completed) or date of last contact (those who discontinued the study early).
Time Frame: From Week 8 to Week 56
Population: The FAS included all randomized subjects who received at least 1 dose of study treatment. Only subjects received study treatment administration at Week 8 are reported.
Measure: Median (95% Confidence Interval); unit: week
Arm/Group | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 50 | 52
week | 37.00 [20.14 to NA] — The upper limit of the 95% confidence interval for the median was not available due to an insufficient number of observed events (ie, the first supplemental aflibercept injections) occurring after the median time point. | 40.79 [20.00 to NA] — The upper limit of the 95% confidence interval for the median was not available due to an insufficient number of observed events (ie, the first supplemental aflibercept injections) occurring after the median time point.

6. Secondary Outcome: Number of Aflibercept Intravitreal Injections up to Week 56 (Including Loading Dose)
Description: Normalized number of aflibercept injections including loading dose was calculated as (number of aflibercept injections received plus all loading doses received) / (time within study period in months), multiplied by 6 months (Week 32) or 12 months (Week 56).
Time Frame: Weeks 32 and 56
Population: The FAS included all randomized subjects who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: normalized no. of aflibercept injections
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 54 | 50 | 52
normalized no. of aflibercept injections
  Week 32 | 3.23 (0.357) | 2.06 (0.583) | 2.13 (0.747)
  Week 56 | 6.33 (0.754) | 3.45 (1.738) | 3.36 (1.854)

7. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness (CST) by Spectral-Domain - Optical Coherence Tomography (SD-OCT) up to Week 56
Description: The SD-OCT assessments in study eye was taken by a study-certified OCT technician according to the standardized procedures described in the Study Manual. Baseline was defined as the last non-missing measurement before the initiation of study treatment.
Time Frame: Baseline (Day 1) and Weeks 32 and 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micron
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 54 | 50 | 52
micron
  Baseline (Day 1) | 265.7 (39.86) | 264.5 (40.26) | 262.9 (34.46)
  Week 32: number analyzed (Participants) | 53 | 48 | 52
  Week 32 | 5.4 (44.52) | 17.8 (42.27) | 10.6 (38.45)
  Week 56: number analyzed (Participants) | 52 | 47 | 52
  Week 56 | 8.1 (58.33) | 12.2 (49.83) | 16.7 (51.98)

8. Secondary Outcome: Change From Baseline in Height of Subretinal Fluid by Spectral-Domain - Optical Coherence Tomography up to Week 56
Description: as for outcome 7
Time Frame: Baseline (Day 1) and Weeks 32 and 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micron
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 54 | 50 | 52
micron
  Baseline (Day 1): number analyzed (Participants) | 30 | 28 | 24
  Baseline (Day 1) | 46.87 (27.753) | 49.84 (32.786) | 50.71 (28.507)
  Week 32: number analyzed (Participants) | 22 | 18 | 17
  Week 32 | 33.05 (62.358) | 18.75 (48.197) | 10.68 (37.686)
  Week 56: number analyzed (Participants) | 23 | 20 | 20
  Week 56 | 22.87 (69.509) | 39.50 (62.183) | 5.95 (38.866)

9. Secondary Outcome: Percentage of Subjects With No Detectable Intraretinal Fluid/Cysts in the Central Subfield up to Week 56
Description: The percentage of subjects with no detectable intraretinal fluid/cysts in the central subfield were summarized by scheduled visit and for any time post-baseline visits. Intraretinal fluid was assessed for the categories 'Absent', 'Present, not clinically significant', 'Present, clinically significant' and 'Not Done'. If intraretinal fluid assessment at any scheduled visit fell under the category 'Absent or Present, not clinically significant', then it was considered as no detectable intraretinal fluid in that scheduled visit.
Time Frame: Weeks 32 and 56
Population: The FAS included all randomized subjects who received at least 1 dose of study treatment. Only subjects analyzed at specific timepoints are reported.
Measure: Number; unit: percentage of subjects
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 53 | 48 | 52
percentage of subjects
  Week 32 | 62.3 | 52.1 | 51.9
  Week 56: number analyzed (Participants) | 52 | 47 | 52
  Week 56 | 59.6 | 59.6 | 51.9

10. Secondary Outcome: Change From Baseline in Total Lesion Area by Fluorescein Angiography (FA) up to Week 56
Description: The total lesion area was defined as the active vascular component [classic and occult choroidal neovascularization (CNV)] and the non-vascular/fibrotic component (fibrosis, serous pigment epithelial detachment, elevated blocking hemorrhage or hyperplastic pigment). Baseline was defined as the last non-missing measurement before the initiation of study treatment.
Time Frame: Baseline (Day 1) and Weeks 32 and 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter square (mm^2)
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 32 | 26 | 26
millimeter square (mm^2)
  Baseline (Day 1) | 5.06884 (4.547571) | 5.48285 (5.488682) | 4.82169 (4.325932)
  Week 32: number analyzed (Participants) | 22 | 19 | 21
  Week 32 | 1.24141 (2.862256) | 1.07111 (2.626369) | 1.13971 (2.024426)
  Week 56: number analyzed (Participants) | 19 | 21 | 18
  Week 56 | 1.56516 (3.226403) | 1.84557 (4.174053) | 2.22914 (3.696873)

11. Secondary Outcome: Change From Baseline in Total Choroidal Neovascularization Area by Fluorescein Angiography up to Week 56
Description: The total CNV area included the measured area of classic and occult components. Baseline was defined as the last non-missing measurement before the initiation of study treatment.
Time Frame: Baseline (Day 1) and Weeks 32 and 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 32 | 26 | 26
mm^2
  Baseline (Day 1) | 5.06 (4.551) | 5.44 (5.531) | 4.77 (4.322)
  Week 32: number analyzed (Participants) | 22 | 19 | 21
  Week 32 | 1.15 (2.968) | 1.10 (2.674) | 1.19 (2.033)
  Week 56: number analyzed (Participants) | 19 | 22 | 18
  Week 56 | 1.46 (3.354) | 1.14 (5.345) | 2.31 (3.656)

12. Secondary Outcome: Systemic Exposure to EYP-1901 Measured Through Plasma Levels up to Week 56
Description: Blood samples were collected at the study visits to determine the EYP-1901 and its main metabolite concentrations.
Time Frame: Up to Week 56
Population: The Pharmacokinetic (PK) set included all subjects in the safety set for whom at least 1 evaluable plasma or aqueous humor (AH) PK sample was available. No subjects were exposed to EYP-1901 in 'Aflibercept 2 mg' reporting group.
Measure: Mean (Standard Deviation); unit: picogram per milliliter
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 0 | 50 | 52
picogram per milliliter
  Week 8 - EYP-1901 concentration: number analyzed (Participants) | 0 | 48 | 51
  Week 8 - EYP-1901 concentration |  | 0.000 (0.0000) | 0.000 (0.0000)
  Week 8 - metabolite concentration: number analyzed (Participants) | 0 | 50 | 51
  Week 8 - metabolite concentration |  | 0.00 (0.00) | 0.00 (0.00)
  Week 20 - EYP-1901 concentration: number analyzed (Participants) | 0 | 46 | 47
  Week 20 - EYP-1901 concentration |  | 23.206 (8.8871) | 27.121 (10.0821)
  Week 20 - metabolite concentration: number analyzed (Participants) | 0 | 46 | 47
  Week 20 - metabolite concentration |  | 1.01 (2.27) | 2.46 (3.86)
  Week 32 - EYP-1901 concentration: number analyzed (Participants) | 0 | 47 | 52
  Week 32 - EYP-1901 concentration |  | 14.333 (6.1098) | 19.335 (7.3783)
  Week 32 - metabolite concentration: number analyzed (Participants) | 0 | 47 | 52
  Week 32 - metabolite concentration |  | 0.00 (0.00) | 0.598 (2.21)
  Week 44 - EYP-1901 concentration: number analyzed (Participants) | 0 | 46 | 51
  Week 44 - EYP-1901 concentration |  | 10.292 (5.2086) | 14.180 (4.9819)
  Week 44 - metabolite concentration: number analyzed (Participants) | 0 | 46 | 51
  Week 44 - metabolite concentration |  | 0.00 (0.00) | 0.485 (1.69)
  Week 56 - EYP-1901 concentration: number analyzed (Participants) | 0 | 45 | 50
  Week 56 - EYP-1901 concentration |  | 7.733 (4.9684) | 10.392 (5.2315)
  Week 56 - metabolite concentration: number analyzed (Participants) | 0 | 45 | 50
  Week 56 - metabolite concentration |  | 0.00 (0.00) | 0.121 (0.867)

13. Secondary Outcome: Ocular Exposure to EYP-1901 Measured Through Aqueous Humor (AH) Levels up to Week 32
Description: The AH samples were collected at the study visits to determine the EYP-1901 and its main metabolite concentrations.
Time Frame: Up to Week 32
Population: The PK set included all subjects in the safety set for whom at least 1 evaluable plasma or AH PK sample was available. No subjects were exposed to EYP-1901 in 'Aflibercept 2 mg' reporting group.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Aflibercept 2 mg | EYP-1901 2060 mcg | EYP-1901 3090 mcg
Number analyzed (Participants) | 0 | 48 | 50
nanogram per milliliter
  Week 8 - EYP-1901 concentration: number analyzed (Participants) | 0 | 46 | 50
  Week 8 - EYP-1901 concentration |  | 0.000 (0.0000) | 0.000 (0.0000)
  Week 8 - metabolite concentration: number analyzed (Participants) | 0 | 43 | 50
  Week 8 - metabolite concentration |  | 0.00 (0.00) | 0.00 (0.00)
  Week 20 - EYP-1901 concentration: number analyzed (Participants) | 0 | 43 | 49
  Week 20 - EYP-1901 concentration |  | 17.426 (13.7143) | 25.066 (18.8594)
  Week 20 - metabolite concentration: number analyzed (Participants) | 0 | 43 | 49
  Week 20 - metabolite concentration |  | 0.00 (0.00) | 0.00 (0.00)
  Week 32 - EYP-1901 concentration |  | 11.890 (10.8436) | 19.813 (15.0833)
  Week 32 - metabolite concentration |  | 0.00 (0.00) | 0.00 (0.00)

14. Secondary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) and Serious Treatment-Emergent Adverse Events up to Week 56
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a patient or clinical investigation subject administered an investigational or marketed (medicinal) product and that does not necessarily have a causal relationship with the product. An serious AE is any AE that results in one of the following outcomes: death; life-threatening; requires in-patient hospitalization; results in a persistent or significant disability/incapacity; congenital anomaly/birth defect; other important medical event. The TEAEs are AEs that occur after the first dose of study treatment.
  administration.
Time Frame: From the study drug administration (Day 1) up to end of the study, approximately 56 weeks.
Population: The Safety analysis set included all subjects who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Aflibercept 2 mg - Study Eye; Aflibercept 2 mg - Systemic: Subjects received aflibercept 2 mg intravitreal injection on Day 1 and at Week 4 followed by intravitreal injection of aflibercept 2 mg and sham injection at Week 8 and then aflibercept 2 mg intravitreal injection once every 8 weeks up to Week 56.
- Aflibercept 2 mg - Fellow Eye; EYP-1901 2060 mcg - Fellow Eye; EYP-1901 3090 mcg - Fellow Eye: No study treatment administered in fellow eye.
- EYP-1901 2060 mcg - Study Eye; EYP-1901 2060 mcg - Systemic: Subjects received aflibercept 2 mg intravitreal injection on Day 1 and at Week 4 followed by intravitreal injection of aflibercept 2 mg and EYP-1901 2060 mcg injection at Week 8 and then intravitreal sham injection once every 8 weeks up to Week 56.
- EYP-1901 3090 mcg - Study Eye; EYP-1901 3090 mcg - Systemic: Subjects received aflibercept 2 mg intravitreal injection on Day 1 and at Week 4 followed by intravitreal injection of aflibercept 2 mg and EYP-1901 3090 mcg injection at Week 8 and then intravitreal sham injection once every 8 weeks up to Week 56.
Arm/Group | Aflibercept 2 mg - Study Eye | Aflibercept 2 mg - Fellow Eye | Aflibercept 2 mg - Systemic | EYP-1901 2060 mcg - Study Eye | EYP-1901 2060 mcg - Fellow Eye | EYP-1901 2060 mcg - Systemic | EYP-1901 3090 mcg - Study Eye | EYP-1901 3090 mcg - Fellow Eye | EYP-1901 3090 mcg - Systemic
Number analyzed (Participants) | 54 | 54 | 54 | 50 | 50 | 50 | 52 | 52 | 52
Participants
  any TEAEs | 30 | 21 | 40 | 30 | 11 | 28 | 30 | 20 | 39
  any Serious TEAEs | 2 | 1 | 6 | 0 | 0 | 6 | 4 | 0 | 9

ADVERSE EVENTS:
Time Frame: TEAEs were collected from the study drug administration (Day 1) up to end of the study, approximately 56 weeks.
Description: The Safety analysis set included all subjects who received at least 1 dose of study treatment.
Arm/Group | Aflibercept 2 mg - Study Eye | Aflibercept 2 mg - Fellow Eye | Aflibercept 2 mg - Systemic | EYP-1901 2060 mcg - Study Eye | EYP-1901 2060 mcg - Fellow Eye | EYP-1901 2060 mcg - Systemic | EYP-1901 3090 mcg - Study Eye | EYP-1901 3090 mcg - Fellow Eye | EYP-1901 3090 mcg - Systemic
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54 | 0/54 | 0/50 | 0/50 | 2/50 | 0/52 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 2/54 | 1/54 | 6/54 | 0/50 | 0/50 | 6/50 | 4/52 | 0/52 | 9/52
Other Adverse Events (participants affected / at risk) | 30/54 | 17/54 | 33/54 | 30/50 | 11/50 | 28/50 | 30/52 | 20/52 | 39/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2 mg - Study Eye (N=54) | Aflibercept 2 mg - Fellow Eye (N=54) | Aflibercept 2 mg - Systemic (N=54) | EYP-1901 2060 mcg - Study Eye (N=50) | EYP-1901 2060 mcg - Fellow Eye (N=50) | EYP-1901 2060 mcg - Systemic (N=50) | EYP-1901 3090 mcg - Study Eye (N=52) | EYP-1901 3090 mcg - Fellow Eye (N=52) | EYP-1901 3090 mcg - Systemic (N=52)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Non-infectious endophthalmitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — This event is not related to study drug or the injection procedure.
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — This event is not related to study drug or the injection procedure.
Vitritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — None of the events were related to study treatment. Events were related to an aflibercept injection and/or paracentesis procedure.
Gastric infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2 mg - Study Eye (N=54) | Aflibercept 2 mg - Fellow Eye (N=54) | Aflibercept 2 mg - Systemic (N=54) | EYP-1901 2060 mcg - Study Eye (N=50) | EYP-1901 2060 mcg - Fellow Eye (N=50) | EYP-1901 2060 mcg - Systemic (N=50) | EYP-1901 3090 mcg - Study Eye (N=52) | EYP-1901 3090 mcg - Fellow Eye (N=52) | EYP-1901 3090 mcg - Systemic (N=52)
Blepharitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 5 (5) | 2 (2) | 0 (0) | 4 (5) | 2 (2) | 0 (0) | 5 (5) | 5 (5) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 4 (8) | 1 (1) | 0 (0) | 6 (7) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Detachment of retinal pigment epithelium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry age-related macular degeneration (Eye disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0)
Retinal oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Subretinal fluid (Eye disorders) | 4 (4) | 0 (0) | 0 (0) | 6 (11) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 8 (8) | 2 (3) | 0 (0) — This event is not related to study drug or the injection procedure.
Vitreous detachment (Eye disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 6 (6) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 4 (5)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 5 (5)
Endophthalmitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — None of the events were related to study treatment. Events were related to an aflibercept injection and/or paracentesis procedure.
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 0 (0) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 4 (4)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 7 (7)

LIMITATIONS AND CAVEATS:
For the events of endophthalmitis in the Serious Adverse Events (SAE) table, none were considered related to EYP-1901. In the aflibercept treatment group, these events were considered related to the injection procedure or were not treatment-related. In the EYP-1901 treatment group, these events were considered related to the supplemental injection procedure (with aflibercept), the paracentesis for aqueous humor collection, or were not treatment-related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT05381948/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT05381948/SAP_001.pdf